CLINICAL TRIAL: NCT02170428
Title: The SKOT I Cohort - a Prospective Cohort Study of Diet and Well-being in Young Danish Children
Brief Title: Diet and Well-being of Young Danish Children
Acronym: SKOT I
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, MD, University of Copenhagen
Other Study IDs: D201; H-KF-2007-0003 (Other: The Committees on Biomedical Research Ethics for the Capital Region of Denmark)
Record Dates: First submitted 2014-06-04; First posted 2014-06-23 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Growth Acceleration; Overweight or Obesity; Biomarkers of Metabolic Syndrome; Programming and Tracking
Keywords: growth,; infancy,; children,; diet,; breastfeeding; complementary feeding; early life programming; tracking; physical activity
MeSH Terms: conditions — Overweight; Obesity; Breast Feeding; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, faeces, white cells, plama/serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- growth and development: Growth and development of a random sample of healthy Danish infants

SUMMARY:
The overall objective with the study was to contribute to the scientific basis for dietary and life strategies, policies and dietary guidelines to infants and young children in Denmark and with special focus on prevention of obesity and diet related chronic diseases such as type 2 diabetes, ischemic heart disease and osteoporosis.

DETAILED DESCRIPTION:
The SKOT I study is a prospective cohort study monitoring healthy young children from 9 to 36 months of age. In 2007, 2211 families from Copenhagen were randomly selected through the National Civil Registry and invited to participate in the study by letter. The participants were invited to three examinations at 9 months ±2 weeks, 18 months ±4 weeks and 36 months ±3 months. A total of 330 children are included in the study, where 312 have completed the 9 months examination, 291 completed the 18 months examination and 263 completed the 3-year examination. All examinations took place at Department of Nutrition, Exercise and Sports, Frederiksberg Denmark. The examinations involved collecting a broad spectrum of data. Following data were collected: anthropometry (weight, height, age- and sex-specific Z-scores for body composition, triceps and subscapularis skinfolds), background interview (concerning e.g. infant feeding, household income, the parent's educational level, allergy and chronic diseases), blood pressure (systolic, diastolic and mean arterial pressure), faeces- and urine sample, blood samples (9 and 36 months), Bio impedance analysis (36 months), 7 day diet registration, general questionaire (concerning e.g. sleep, daycare, attendance and use of screen devices), psychomotor questionnaire (motoric development), 7 day physical activity monitoring and dual energy x-ray absorptiometry scan (36 months).

ELIGIBILITY:
Inclusion Criteria:

* healthy singletons born at term (week 37-43) between August 2006 and September 2007 with no disease that could influence food intake or growth

Exclusion Criteria:

* born preterm (before week 37)
* non-Danish speaking parents.

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy young Danish Children selected through the National Civil Registry and invited to participate by letter.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in anthropometric measurements in periods of early childhood. | 9, 18 and 36 months of age
  Composite outcome consisting of body weight, height, body mass index (BMI) and BMI z-scores, waist-, upper arm- and head circumference, skinfold thickness measured at subscapularis and triceps.
Body composition in early childhood | 36 months of age
  Body composition is measures by Dual-energy X-ray Absorptiometry and bio impedance. Fat mass, fat mass index (kg/m2), fat free mass index (kg/m2) are calculated.
Metabolic syndrome score in early life | 9 and 36 months of age
  Composite outcome consisting of triglycerides, high lipoprotein (HDL) and glucose measured in plasma/serum, waist circumference and blood pressure.
Diet in periods of early life | 9, 18 and 36 months of age
  The diet is recorded using self-reported 7-day record questionnaire.

SECONDARY OUTCOMES:
Breastfeeding duration in infancy and early childhood | 9, 18 and 36 months of age
  Questionnaire used for assessment of exclusive and partially breastfeeding.
Insulin like growth factor at 9 and 36 months of age | 9 and 36 months of age
  Insulin like growth factor-1 and insulin like growth factor binding protein-3 concentrations in plasma.
Physical activity, sedentary behavior and sleep in early childhood | 9, 18 and 36 months of age
  Physical activity and sedentary behavior measured by ActiGrafph GT3X accelerometer, recording for 24 hours in 7 days at 36 months of age. Information on outdoor activity, sedentary behavior and night sleep are collected through questionnaires at 9, 18 and 36 months of age.
Bone mass in 3-year-old children | 36 months of age
  Bone mass is measured by Dual-energy X-ray Absorptiometry
Vitamin D status in infancy | 9 months of age
  25-hydroxyvitamin D concentrations are analysed in blood samples at 9 months of age.
Allergy and chronic diseases | 9 and 36 months of age
  Assessment of diseases by questionnaires
Appetite hormones in infancy | 9 months of age
  Leptin and adiponectin concentrations measured from blood samples
Change in gut microbiota | 9, 18 and 36 months of age
  Microbiota in the faeces analysed using polymerase chain reaction (PCR)
Achievement of milestones | 9 and 36 months of age
  Achievement of age-specific milestones by questionnaires; WHO questionnaires at 9 and 36 months of age and Ages & Stages Questionnaires (ASQ) at 36 months of age
Metabolomics in the urine | 9, 18 and 36 months of age
  Metabolomics analysed using urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, MD Professor, Principal Investigator — Faculty of Science, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Sciences, University of Copenhagen, Frederiksberg, Denmark